CLINICAL TRIAL: NCT05022589
Title: Remote Digital Health Intervention to Improve Balance and Reduce Fall Risk
Acronym: rSTAND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Posit Science Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PSC-0820-21
Record Dates: First submitted 2021-08-20; First posted 2021-08-26 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Fall

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Treatment (Experimental): Computerized plasticity-based adaptive cognitive training requiring a total maximum of 50 treatment sessions, 5 sessions per week, ~30 minutes per session.
  Interventions: Other: Computerized Plasticity-Based Adaptive Cognitive Training

INTERVENTIONS:
Other: Computerized Plasticity-Based Adaptive Cognitive Training — Computerized plasticity-based adaptive cognitive training requiring a total maximum of 50 treatment sessions, 5 sessions per week, ~30 minutes per session.
  Other Names: rSTAND

SUMMARY:
The goal of this project is to further develop and evaluate a computerized cognitive-training program designed to extend older adults' functional independence and reduce accidental falls (i.e., reduce factors that contribute to fall risk; including cognitive abilities/executive functions). This intervention may benefit a large population of vulnerable older adults with elevated fall risk and lack of long-term viable treatment options.

DETAILED DESCRIPTION:
The investigators will employ a single arm study open label usability/feasibility study comprised of a computerized training program that targets core executive functions (working memory, inhibition), speed of processing and sustained attention, and is grounded on design principles that drive adaptive brain plasticity to improve cognitive function and bolster functional abilities in older adults with an elevated fall risk.

ELIGIBILITY:
Inclusion Criteria:

1. Participants who are 65 years of age or older.
2. Participants must be US residents.
3. Participant with at least one self-reported fall within the last 1 year or difficulty walking one half a mile or difficulty climbing one flight of stairs.
4. Participants who are fluent English speakers from the age of 12, per self-report, to ensure reasonable neuropsychological results on key assessments.
5. Participant must have adequate sensorimotor capacity to perform the program, including visual capacity adequate to read from a computer screen at a normal viewing distance, auditory capacity adequate to understand normal speech, and motor capacity adequate to control a computer mouse or a tablet.

Exclusion Criteria:

1. Participants had joint replacement surgery or significant join/leg injury less than one year prior to the screening visit.
2. Participants have a joint replacement surgery scheduled within the next 6 months.
3. Participants use a walker or wheelchair on a regular basis.
4. Participants have a diagnosis of benign paroxysmal positional vertigo (BPPV), labyrinthitis or suffers migraines that result in chronic vertigo.
5. Participants self-reports vision or hearing difficulties that would interfere with the ability to complete the study tasks.
6. Participants with untreated psychiatric conditions, including substance abuse/dependence disorders, recent hospitalization, ongoing chemotherapy or other cancer treatment.
7. Participants with medical illnesses, injuries or conditions predisposing to imminent functional and/or cognitive decline (e.g. multiple sclerosis, stroke, traumatic brain injury, dementia, etc.)
8. Participants enrolled in a concurrent clinical trial involving an intervention targeting physical functioning to prevent falls; investigational pharmaceutical; nutraceutical; medical device; or behavioral treatment that could affect the outcome of this study. However, participation in standard treatments (e.g., occupational therapy) or use of prescribed medications (e.g., anti-depressants) is allowable.
9. Participants using computer-based cognitive training programs or has used it within a month of the consent date.
10. Participants who answered 'yes' to questions 4 (Active Suicidal Ideation with Intent) or 5 (Active Suicidal Ideation with Specific Plan and Intent) on the Columbia-Suicide Severity Rating Scale (C-SSRS) or 'yes' to any of the suicide-related behaviors (actual attempt, interrupted attempt, aborted attempt, preparatory act or behavior) on the C-SSRS "Suicidal Behavior" if the ideation or behavior occurred within 2 months from Participant's date of consent.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 23 (Actual)
Dates: Start 2022-08-09 (Actual); Primary Completion 2024-04-19 (Actual); Study Completion 2024-04-19 (Actual)

PRIMARY OUTCOMES:
Net Promoter Score | At 10 weeks
  The scoring for this answer is based on a 0 to 10 scale. Those who respond with a score of 9 to 10 are called Promoters, and are considered likely to exhibit value-creating behaviors, such as making more positive referrals to other potential program participants. Those who respond with a score of 0 to 6 are labeled Detractors, and they are believed to be less likely to exhibit the value-creating behaviors. Responses of 7 and 8 are labeled Passives, and their behavior falls between Promoters and Detractors. The Net Promoter Score is calculated by subtracting the percentage of customers who are Detractors from the percentage of customers who are Promoters. For purposes of calculating a Net Promoter Score, Passives count toward the total number of respondents, thus decreasing the percentage of detractors and promoters and pushing the net score toward 0.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Van Vleet, PhD, Principal Investigator — Posit Science Corporation
Locations (1):
- Posit Science Corporation, San Francisco, California, United States